CLINICAL TRIAL: NCT06212310
Title: Genetic Counseling Service Delivery and Outcomes in Diverse and Underserved Populations
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Society of Genetic Counselors (Other)
Responsible Party: Principal Investigator, Sara Pirzadeh-Miller, Associate Director, Cancer Genetics Program, University of Texas Southwestern Medical Center
Other Study IDs: 2021-1008
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Genetic Predisposition
Keywords: genetic counseling service delivery
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In-person genetic counseling: Patients referred for standard of cancer genetic counseling are seen in-person with a genetic counselor for service.
- Telephone genetic counseling: Patients referred for standard of cancer genetic counseling are on the telephone with a genetic counselor for service.

SUMMARY:
This 2-arm prospective, randomized, controlled clinical trial compared outcomes of telephone genetic counseling (intervention) versus in-person genetic counseling (control) in an underserved, multilingual patient population referred for cancer genetic counseling at two North Texas safety-net hospitals.

The main question[s] it aims to answer are:

* Is telephone genetic counseling equal to in-person genetic counseling in the patient reported outcomes? Cancer genetics knowledge, attitude towards GT, and informed choice as well as GC-specific empowerment.
* Is telephone genetic counseling-based clinical outcomes the same as in-person genetic counseling for visit completion and testing rates? Participants will be randomized to either in-person or telephone genetic counseling arm and complete standard of care genetic counseling visit process where testing is offered. Both arms will complete a series of surveys to assess the outcomes of interest.

DETAILED DESCRIPTION:
The overarching goal of this pilot prospective randomized controlled study is to compare patient-reported and clinical operations outcomes between in-person genetic counseling (IPGC - control) and telephone-based genetic counseling (TGC - intervention) in an indigent English or Spanish-speaking population seeking genetic counseling for hereditary cancer syndromes to create a framework for effective and efficient genetic service delivery in these populations nationally. General genetic education and principles will be conveyed through a standard genetic counseling session including a pre-test education video in both the TGC and IPGC arms. The primary project objectives are to compare the following outcomes between the IPGC and TGC study arms. Aim 1: Patient reported outcomes - A. Patient satisfaction with genetic counseling visit; B. Knowledge of basic principles of cancer genetics and implications of genetic testing for personal healthcare and relatives. Secondary objectives for this aim are: 1. Patient ability to make informed choice; and 2. Genetic counseling-specific empowerment outcomes. Aim 2: Clinical outcomes - visit completion rate; Secondary objectives are: 1. Genetic testing completion rate; and 2. Genetic testing cancelation/failure rate. Investigators hypothesize that patients in the TGC arm will not have significant differences in knowledge, satisfaction, informed choice or genetic counseling-specific empowerment compared to the IPGC arm. Investigators also expect significantly increased visit completion rate and lower test completion rate in the TGC arm compared to the IPGC arm, but no significant difference in sample failure rate.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Patients who are English or Spanish-speaking
* Adults (18 years and older)
* Patients scheduled for cancer genetic counseling
* Patients must either be uninsured or have Medicaid
* Patients must have no prior germline genetic testing or cancer genetic counseling
* Patients must have a working telephone number and valid e-mail address
* Patients must have Internet access to complete electronic study surveys, and receive study-related documents electronically

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals referred to genetic counseling as part of standard of care
Sampling Method: Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pirzadeh-Miller, M.S., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2022 and 2023, adult patients referred for cancer genetic counseling at two cancer genetics clinics housed in two safety-net hospitals in North Texas were recruited for the study. Patients had to meet the following inclusion criteria: be age 18 or older; speak English or Spanish; be uninsured or have Medicaid; have no prior cancer genetic counseling or testing; and have internet access, a valid email, and a working telephone number. Patients were excluded if they met exclusion criteria.
Pre-assignment Details: Vulnerable populations and patients referred to genetic counseling for surgical planning were excluded from the study and were not assigned to a study arm.
Groups:
- Telephone Genetic Counseling: Patients referred for standard of cancer genetic counseling are on the telephone with a genetic counselor for service.
  Telephone genetic counseling: genetic counseling service delivered audio-only
Period: Overall Study
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling
Started | 212 | 207
Completed | 100 | 101
Not Completed | 112 | 106

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 100 | 198
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 92 | 181
  Male | 11 | 9 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — American Indian or Alaska Native; Asian; Black or African American; White, Hispanic or Latino; White, Non-Hispanic or Latino; Hispanic or Latino, NOS
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 1 | 0 | 1
    White, Hispanic or Latino | 42 | 44 | 86
    White, Non-Hispanic or Latino | 11 | 13 | 24
    Hispanic or Latino, NOS | 33 | 21 | 54
    Black or African American | 13 | 22 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 101 | 201
Preferred Language [Count of Participants; unit: Participants] — Participant-reported preferred language (English, Spanish)
  Participants
    English | 47 | 55 | 102
    Spanish | 53 | 46 | 99
Cancer Diagnosis [Count of Participants; unit: Participants] — Participant-reported personal history of cancer diagnosis (Yes, No)
  Participants
    Yes | 35 | 23 | 58
    No | 65 | 78 | 143

OUTCOME MEASURES:

1. Primary Outcome: Change in Knowledge Score
Description: Measure change in knowledge of basic principles of cancer genetics and implications of genetic testing for personal healthcare and relatives pre- and post- genetic counseling using the Multi-dimensional Model of Informed Choice (MMIC) scale knowledge score, with minimum and maximum scores of 0 and 8 respectively, and higher scores correlated with better knowledge
Time Frame: MMIC Survey administered within 7 days prior to and post-genetic counseling visit
Population: Population who completed genetic counseling and all study surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling
Number analyzed (Participants) | 100 | 101
score on a scale | 0.05 (1.37) | -0.08 (1.51)

2. Primary Outcome: Patient Reported Outcome of Patient Satisfaction
Description: Measure patient-reported patient satisfaction with genetic counseling visit using the Genetic Counseling Satisfaction Scale (GCSS) scores, with minimum and maximum values of 6 and 30 respectively and higher scores correlated with higher satisfaction
Time Frame: GCSS survey administered within 7 days post-genetic counseling visit
Population: Participants who completed genetic counseling and all study surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling
Number analyzed (Participants) | 100 | 101
score on a scale | 24.64 (5.38) | 25.27 (3.75)

3. Primary Outcome: Clinical Outcome Measure of Genetic Counseling Visit Completion
Description: Measure difference in genetic counseling visit completion rate between study arms
Time Frame: Genetic counseling visit completion was evaluated daily, up to 13.5 months
Population: Participants who completed the Pre-Genetic Counseling Survey and were scheduled for genetic counseling (in-person or via telephone) through the study
Measure: Count of Participants; unit: Participants
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling
Number analyzed (Participants) | 171 | 146
Participants | 141 | 131

4. Secondary Outcome: Patient Reported Outcome of Genetic Counseling-specific Empowerment
Description: Measure change in patient reported genetic counseling-specific empowerment pre and post-genetic counseling using the Genomic Outcome Scale (GOS) scores with minimum and maximum scores of 6 and 30 respectively and higher scores correlated with improved outcomes
Time Frame: GOS survey administered within 7 days prior to and post-genetic counseling visit
Population: Participants who completed genetic counseling and all study surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling
Number analyzed (Participants) | 100 | 101
score on a scale | -0.21 (5.34) | 0.86 (4.62)

5. Secondary Outcome: Number of Participants That Made an Informed Choice
Description: Participants' ability to make an informed choice is assessed by the number of participants that made an informed choice using the Multi-dimensional Model of Informed Choice composite tool that includes understanding of relevant knowledge (1-8 items-higher scores indicate greater knowledge), attitudes toward testing (1-5 items-higher scores represent more positive attitudes), and whether the test decision is congruent with personal values (positive or negative about testing in relation to whether testing was accepted or declined).
Time Frame: MMIC survey administered within 7 days post-genetic counseling and genetic testing uptake during scheduled genetic counseling appointment
Population: Participants who completed genetic counseling and all study surveys
Measure: Count of Participants; unit: Participants
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling
Number analyzed (Participants) | 100 | 101
Participants | 39 | 53

6. Secondary Outcome: Clinical Outcome Measure of Genetic Testing Completion
Description: Measure genetic test completion rate between study arms
Time Frame: Sample for testing provided within 45 days of visit without sample failure
Population: Sample failures/test cancellations amongst participants who elected genetic testing
Measure: Count of Participants; unit: Participants
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling
Number analyzed (Participants) | 86 | 81
Participants
  Blood sample; completed genetic test | 83 | 20
  Blood sample; incomplete genetic test | 0 | 3
  Saliva sample; completed genetic test | 3 | 40
  Saliva sample; incomplete genetic test | 0 | 18

ADVERSE EVENTS:
Time Frame: This was a minimal risk study and adverse events data were not collected
Description: Adverse Events not monitored/assessed. This was a minimal risk study.
Arm/Group | In-person Genetic Counseling | Telephone Genetic Counseling
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Use of non-validated instruments (Multi-dimensional Model of Informed Choice and Genomics Outcome Scale), higher drop-off rate of enrolled study participants (50% observed; 30% anticipated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT06212310/Prot_SAP_000.pdf